CLINICAL TRIAL: NCT02278913
Title: Basal Bolus Regimen With Insulin Analogs Versus Human Insulin in Medical Patients With Type 2 Diabetes: A Randomized Controlled Trial in Paraguay
Brief Title: Basal Bolus Versus Human Insulin in Hospitalized Patients With Diabetes in Paraguay
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Universidad Nacional de Asunción (Other)
Responsible Party: Principal Investigator, Elvio Dario Bueno Colman, Jefe de Departamento de Endocrinologia y Diabetes, Hospital de Clínicas, Universidad Nacional de Asunción-Paraguay (U.N.A)., Universidad Nacional de Asunción
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P 08/09
Record Dates: First submitted 2014-10-24; First posted 2014-10-30 (Estimated); Last update posted 2014-10-30 (Estimated); Status verified 2014-10

CONDITIONS: Hyperglycemia; Diabetes
Keywords: inpatient; hospital; randomized trial; diabetes; analogs; human insulin
MeSH Terms: conditions — Hyperglycemia; Diabetes Mellitus; Insulin Resistance | interventions — Insulin Glargine; Insulin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Basal Bolus (Glargine and Glulisine) (Experimental): Basal bolus: with Insulin analogs (glargine and glulisine), 50% of total daily dose as glargine given before breakfast and 50% as glulisine insulin given in three equally divided doses before each meal.
  Interventions: Drug: Basal Bolus (Glargine and Glulisine)
- Human Insulin (Active Comparator): Human insulin: NPH and regular insulin: 2/3 of total daily dose as NPH and 1/3 as regular insulin. NPH insulin dose given as 2/3 in the morning before breakfast and 1/3 before dinner. Regular insulin given in three equally divided doses before each meal
  Interventions: Drug: Human Insulin

INTERVENTIONS:
Drug: Basal Bolus (Glargine and Glulisine) — Glargine daily + Glulisine before meals
  Other Names: Glargine and glulisine
  Arms: Basal Bolus (Glargine and Glulisine)
Drug: Human Insulin — NPH twice a day + Regular insulin before meals
  Other Names: NPH and regular
  Arms: Human Insulin

SUMMARY:
Few randomized studies have focused on the optimal management of non-ICU patients with type 2 diabetes in Latin America. Objective: Compare safety and efficacy of a basal bolus regimen with analogs and human insulins in general medicine patients admitted to a University Hospital in Asuncion, Paraguay.

DETAILED DESCRIPTION:
Few randomized intervention inpatient trials have been conducted in Latin America to determine optimal treatment regimens for patients with type 2 diabetes. In the absence of regional guidelines, most international societies in Latin America recommend following international guidelines for the management of hospitalized patients with diabetes. However, hospital resources, admission cause and inpatient glycemic control differ among countries. In the US, the leading cause of admission to the hospital in patients with diabetes is cardiovascular disease, whereas infections and acute complications of diabetes are more common than cardiovascular disease in some countries. The safety and efficacy of insulin regimens in non-ICU setting in Latin countries have not been determined. Objective: to compare the efficacy and safety of a basal-bolus regimen using insulin analogs with glargine once daily plus glulisine before meals to human insulin with NPH twice daily and regular insulin before meals in medicine patients with type 2 diabetes Outcome measures. To determine differences in glycemic control between groups as measured by mean daily BG concentration during the hospital stay. Secondary outcomes included differences between treatment groups in any of the following measures: number of hypoglycemic events (BG <70 mg/dL and <40 mg/dL), total daily dose of insulin, length of hospital stay, hospital complications and mortality.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years
* History of type 2 diabetes > 1 month
* Treatment with diet alone, any combination of oral antidiabetic agents, and/or insulin prior to admission
* Absence of diabetic ketoacidosis

Exclusion Criteria:

* No history of diabetes
* Subjects expected to undergo surgery during the hospitalization course
* Clinically relevant hepatic disease
* Impaired renal function (serum creatinine ≥ 3.0 mg/dL)
* Pregnancy
* Any mental condition rendering the subject unable to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 134 (Actual)
Dates: Start 2009-04; Primary Completion 2010-04 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Glycemic control | During hospitalization, an expected average of 10 days
  The primary outcome of the study is to determine differences in glycemic control as measured by mean daily BG concentration between human insulin (NPH + Regular insulin) and basal bolus therapy (glargine once daily + glulisine)

SECONDARY OUTCOMES:
Hypoglycemia | During hospitalization, an expected average of 10 days
  Number of hypoglycemic events (<70 mg/dl) and severe hypoglycemic events (<40 mg/dl)
Insulin dose | During hospitalization, an expected average of 10 days
  Total daily dose of insulin
Length of stay | During hospitalization, an expected average of 10 days
  Duration of hospitalization
Mortality | During hospitalization, an expected average of 10 days
  Mortality is defined as death occurring during admission

CONTACTS AND LOCATIONS:
Overall Officials: Elvio Bueno, MD, Principal Investigator — Universida Nacional de Asuncion
Locations (1):
- Clínica Médica del Hospital de Clínicas, Universidad Nacional de Asunción,, Asunción, Paraguay